CLINICAL TRIAL: NCT04205006
Title: Long-term Outcome of a Pragmatic Trial of Multifaceted Intervention (STROKE-CARD Care) to Reduce Cardiovascular Risk and Improve Quality-of-life After Ischemic Stroke and Transient Ischemic Attack
Brief Title: Stroke Card Long-term Follow-Up
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Medical University Innsbruck (Other)
Collaborators: VASCage GmbH (Other); Tirol Kiniken GmbH (Other); Barmherzige Brüder Vienna (Other)
Responsible Party: Sponsor
Other Study IDs: SCFU
Record Dates: First submitted 2019-12-13; First posted 2019-12-19 (Actual); Last update posted 2022-08-30 (Actual); Status verified 2022-04

CONDITIONS: Ischemic Stroke; TIA
Keywords: ischemic stroke; secondary prevention; transient ischemic attack; disease management
MeSH Terms: conditions — Ischemic Stroke; Ischemic Attack, Transient

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum and whole blood sample.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- STROKE CARD Cohort: Consecutive patients treated at the Department of Neurology of the University Hospital Innsbruck with ischemic stroke or high-risk TIA between 2013 and 2018 and enrolled in the Stroke Card trial, (except for those who aborted the previous trial).

SUMMARY:
We undertook the STROKE-CARD trial (NCT02156778) between 2014 and 2018 with follow-up until 2019 to evaluate the efficacy of the Post-Stroke disease-management program STROKE-CARD care. To further investigate the long-term efficacy of STROKE-CARD care all participants of the original trial will be invited for a Long-term in Person follow-up (3 - 6 years).

ELIGIBILITY:
Inclusion Criteria:

* Inclusion in the previous STROKE-CARD trial (NCT02156778)
* Written informed consent

Exclusion Criteria:

* none

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients from the STROKE-CARD trial (n=2149) will be contacted by phone or mail for possible enrolment in the study. The STROKE-CARD cohort included consecutive patients with acute ischaemic stroke or TIA (ABCD2-Score ≥ 3) admitted to one of the two study centres (Medical University of Innsbruck, Hospital St. John's of God Vienna) between 2014 and 2018.
Sampling Method: Non-Probability Sample
Enrollment: 1000 (Estimated)
Dates: Start 2019-12-16 (Actual); Primary Completion 2022-11-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
The composite CVD outcome: nonfatal stroke (ischemic or hemorrhagic) | through study completion, an average of 4,5 years
  Recurrent stroke
The composite CVD outcome: nonfatal myocardial infarction | through study completion, an average of 4,5 years
  Major recurrent (post-discharge) cardiac event
The composite CVD outcome: vascular death | through study completion, an average of 4,5 years
  death resulting from an acute myocardial infarction, sudden cardiac death, death due to heart failure, stroke, cardiovascular procedures, and death due to other CV causes.
self-reported health-related quality of life | through study completion, an average of 4,5 years
  quantified with the European Quality of Life 5-Dimensions 3-Levels (EQ-5D-3L) overall health utility score14 with rescaled European visual analogue scale weights.

SECONDARY OUTCOMES:
The composite outcome of stroke/TIA | through study completion, an average of 4,5 years
  TIA defined as transient neurological deficit <24h and absence of DWI positive lesions on MRI
all-cause mortality | through study completion at long term follow up visit, an average of 4,5 years
  death from all causes
EQ-ED-3L | through study completion at long term follow up visit, an average of 4,5 years
  individual 3-level components of the European Quality of Life 5-Dimensions 3-Levels (EQ-5D-3L) questionnaire14 (i.e. mobility, self-care, usual activities, no pain or discomfort, no anxiety or depression) comparing people reporting no problems (level 1) with those reporting problems (level 2 and 3)
Proportions of participants achieving target levels of risk factors in each trial arm of the previous STROKE-CARD trial. | through study completion at long term follow up visit, an average of 4,5 years
  Blood pressure <140/<90 mmHg or <130/<85 mmHg in patients with diabetes mellitus, severe renal impairment; HbA1c <7.5% at the study visit in patients with diabetes mellitus; having quit smoking by the study visit in patients that had been smokers at baseline in the STROKE-CARD trial; LDL cholesterol < 100 mg/dL or <70 mg/dL in high-risk patients (i.e. stroke or TIA due to large-artery atherosclerosis or small-vessel occlusion, other evidence of atherosclerotic vascular disease, baseline diabetes; Metabolic Syndrome (NCEP-ATPIII): reduction of component number by 1, physical activity >90 minutes; Platelet inhibitor or oral anticoagulation; Oral anticoagulation (INR 2-3, Time in Therapeutic Range (TTR)>70%) in case of atrial fibrillation (AF), Lipid-lowering medication except for non-atherosclerotic strokes (e.g. vessel dissection).

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Kiechl, Prof. Dr., Principal Investigator — Medical University of Innsbruck, Austria, Department of Neurology; Wilfried Lang, Prof. Dr., Principal Investigator — Hospital St. John's of God, Vienna, Austria, Department of Neurology
Locations (2):
- Austria (2):
  - Medical University of Innsbruck, Department of Neurology, Innsbruck, Tyrol
  - Hospital St. John's of God, Vienna

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Toell T, Boehme C, Mayer L, Krebs S, Lang C, Willeit K, Prantl B, Knoflach M, Rumpold G, Schoenherr G, Griesmacher A, Willeit P, Ferrari J, Lang W, Kiechl S, Willeit J. Pragmatic trial of multifaceted intervention (STROKE-CARD care) to reduce cardiovascular risk and improve quality-of-life after ischaemic stroke and transient ischaemic attack -study protocol. BMC Neurol. 2018 Nov 6;18(1):187. doi: 10.1186/s12883-018-1185-2. PMID 30400876
- [Result] Boehme C, Toell T, Mayer-Suess L, Domig L, Pechlaner R, Willeit K, Tschiderer L, Seekircher L, Willeit P, Griesmacher A, Knoflach M, Willeit J, Kiechl S. The dimension of preventable stroke in a large representative patient cohort. Neurology. 2019 Dec 3;93(23):e2121-e2132. doi: 10.1212/WNL.0000000000008573. Epub 2019 Oct 31. PMID 31672716
- [Derived] Karisik A, Dejakum B, Moelgg K, Granna J, Felicetti S, Pechlaner R, Mayer-Suess L, Toell T, Buergi L, Scherer L, Willeit K, Heidinger M, Lang C, Ferrari J, Krebs S, Kleyhons R, Resch H, Willeit J, Seekircher L, Tschiderer L, Willeit P, Sykora M, Schett G, Lang W, Knoflach M, Kiechl S, Boehme C. Incidence, characteristics, and consequences of fractures after acute ischemic stroke and TIA-A prospective cohort study. Int J Stroke. 2025 Oct;20(9):1141-1149. doi: 10.1177/17474930251345300. Epub 2025 May 20. PMID 40391684
- [Derived] Boehme C, Domig L, Komarek S, Toell T, Mayer L, Dejakum B, Krebs S, Pechlaner R, Bernegger A, Mueller C, Rumpold G, Griesmacher A, Vigl M, Schoenherr G, Schmidauer C, Ferrari J, Lang W, Knoflach M, Kiechl S. Long-term outcome of a pragmatic trial of multifaceted intervention (STROKE-CARD care) to reduce cardiovascular risk and improve quality-of-life after ischaemic stroke and transient ischaemic attack: study protocol. BMC Cardiovasc Disord. 2022 Aug 1;22(1):347. doi: 10.1186/s12872-022-02785-5. PMID 35915405